CLINICAL TRIAL: NCT00146419
Title: Study to Understand the Natural History of HIV/AIDS in the Era of Effective Therapy (SUN Study)
Status: Completed | Type: Observational
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: The Miriam Hospital (Other); Hennepin Healthcare Research Institute (Other); Washington University School of Medicine (Other); Denver Infectious Disease Consultants, PLLC (Other)
Responsible Party: Sponsor
Other Study IDs: CDC-NCHSTP-3979; 200-2002-00610; 200-2002-00611; 200-2002-00612; 200-2002-00613
Record Dates: First submitted 2005-09-01; First posted 2005-09-07 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2012-09

CONDITIONS: HIV Infections; Sexually Transmitted Diseases
Keywords: Treatment Experienced; Treatment Naive
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Reduction in behaviors capable of sexually transmitting HIV — Clinic-level risk reduction counseling

SUMMARY:
The SUN Study is a Centers for Disease Control and Prevention (CDC)-sponsored multi-site prospective observational cohort study designed to better understand the incidence and etiology of metabolic and other complications related to effective HIV treatment and longer survival. The SUN Study is also providing a platform to evaluate a behavioral intervention designed to reduce HIV transmission through prevention counseling in routine care.

DETAILED DESCRIPTION:
Effective antiretroviral therapy has significantly improved and prolonged the lives of HIV-infected persons. However, antiretroviral use has also been associated with a diverse array of "unnatural" metabolic complications and other adverse medical conditions. These problems, together with subsequent longer survival, have increased patients' risk for developing renal, hepatic, cardiovascular, neurological, rheumatologic, and other end-organ diseases, and cancers. Longer survival is also increasing the pool of HIV-infected persons capable of transmitting the virus, which could accelerate the pace of the U.S. epidemic; however, the ability of physicians caring for HIV-infected persons to incorporate prevention into their clinical practices and the effectiveness of this intervention have not been extensively evaluated.

The goals of the Study to Understand the Natural History of HIV and AIDS ("SUN" Study) are:

* to monitor the incidence of metabolic and other medical complications related to the treatment of HIV infection and attendant prolonged survival,
* to identify risk factors associated with the development of these metabolic and other medical complications,
* to monitor the contribution of these complications and other conditions to the morbidity and mortality of HIV infection, and
* to evaluate the efficacy of a structured program of prevention activities, which are integrated into the routine medical care of HIV patients to reduce HIV transmission.

The SUN Study is designed to enroll and follow for 5 or more years a cohort of up to 1,000 HIV-infected adults at HIV specialty care centers in four U.S. cities: Denver, Minneapolis, Providence, and St. Louis. Data will be gathered through longitudinal real-time chart review, biannual physical examination (e.g., body mass index [BMI], blood pressure), repeated non-invasive imaging (e.g., dual energy x-ray absortiometry [DEXA] scanning, carotid ultrasonography) and regularly scheduled laboratory testing (e.g., serum lipids, pap smears, and urinary microalbumin). Data collection and quality control will be managed by Cerner Corporation. After sufficient enrollment, (circa 200 persons per site) a structured prevention program to reduce HIV transmission will be introduced. The impact of this intervention will be evaluated both subjectively (e.g., self-reported change in behavior on an audio computer-assisted self-interviewing [ACASI] questionnaire) and objectively (e.g., change in sexually transmitted disease [STD] incidence).

Outcomes include determination of the incidence of therapy-related metabolic complications and other adverse conditions associated with longer survival, identification of risk factors for these complications and conditions, and reduction in both reported and objective measures of risky sexual behavior.

ELIGIBILITY:
Inclusion Criteria:

* Subject is age 18 years or older.
* Subject is HIV-infected as confirmed by positive enzyme immunoassay (EIA) and western blot testing, by an HIV viral load >5,000 copies, or by genotyping that confirms infection with HIV.
* For highly active antiretroviral therapy (HAART)-naïve subjects (i.e. persons with no prior substantial antiretroviral [ARV] exposure):

  * Subject's CD4+ cell count is between 100 and 500 cells/mm³
  * Subject has not ever received more than 30 days consecutive or non-consecutive treatment with any ARVs regardless of reason (e.g., pharmacokinetic study, post-exposure prophylaxis, prevention of vertical transmission in pregnancy).
* For HAART-exposed subjects (i.e. persons who have taken or are taking HAART at the time of enrollment):

  * Subject's CD4+ cell count is >100 cells/mm³
  * Subject's previous and/or current treatment with ARVs has consisted only of HAART (of any duration and in any number of regimens) defined as:

    * >3 antiretroviral drugs from at least 2 antiretroviral drug classes (nucleotide reverse transcriptase inhibitors [NRTI], non-nucleoside reverse transcriptase inhibitors [NNRTI], protease inhibitors [PI]); or,
    * >3 NRTIs.
* Other antiretroviral combinations that in the course of the study are developed and become accepted as equivalent to best available therapy.
* Subject has received only HAART either as prescribed therapy or in the context of a supervised study.
* Subject has completed at least two visits within the past year to the clinical facility where the patient is eligible for enrollment.
* Subject is anticipated to continue receiving care at the clinical facility where she or he is eligible for enrollment for at least 2 years.
* Subject is able to understand and sign an informed consent.

Exclusion Criteria:

* Subject is pregnant.
* Subject is incarcerated. (footnote 1)
* Within the past 60 days subject has:

  * Had an AIDS-defining opportunistic infection or illness.
  * Received any chemotherapy or immunomodulating therapy (e.g., glucocorticoids, interleukin-2, interferon). (footnote 2)
* Subject is expected to live less than 2 years.
* Subject is unable or unwilling to complete any part of the study protocol.
* Subject is considered by the principal investigator to be ineligible for enrollment for any other reason, including but not limited to remote geographic location, experience in prior research studies, inconsistency as a historian, etc.
* Subject is unable or refuses to provide informed written consent due to any physical or psychological incapacity (e.g., persistent vegetative state, mental disability).

Footnotes:

1. Participants will be temporarily suspended from the study while pregnant or incarcerated after enrollment.
2. Cases where eligibility by these criteria is unclear or requires special consideration will be referred to the Executive Committee for a final decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV-infected persons receiving care at HIV-specialty clinics
Sampling Method: Non-Probability Sample
Enrollment: 699 (Actual)
Dates: Start 2004-03; Primary Completion 2006-08 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Carpenter, M.D., Principal Investigator — The Miriam Hospital; Keith Henry, M.D., Principal Investigator — Hennepin Healthcare Research Institute; Kristin Mondy, M.D., Principal Investigator — Washington University School of Medicine; John H Hammer, M.D., Principal Investigator — Denver Infectious Disease Consultants, PLLC
Locations (8):
- United States (8):
  - Denver Infectious Disease Consultants, Denver, Colorado
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Park-Nicollet Institute, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - The Miriam Hospital, Providence, Rhode Island
  - Cerner Corporation, McLean, Virginia

REFERENCES:
- [Background] Vellozzi C, Brooks JT, Bush TJ, Conley LJ, Henry K, Carpenter CC, Overton ET, Hammer J, Wood K, Holmberg SD; SUN Study Investigators. The study to understand the natural history of HIV and AIDS in the era of effective therapy (SUN Study). Am J Epidemiol. 2009 Mar 1;169(5):642-52. doi: 10.1093/aje/kwn361. Epub 2008 Dec 13. PMID 19074775
- [Background] Kojic EM, Cu-Uvin S, Conley L, Bush T, Onyekwuluje J, Swan DC, Unger ER, Henry K, Hammer JH, Overton ET, Darragh TM, Palefsky JM, Vellozzi C, Patel P, Brooks JT. Human papillomavirus infection and cytologic abnormalities of the anus and cervix among HIV-infected women in the study to understand the natural history of HIV/AIDS in the era of effective therapy (the SUN study). Sex Transm Dis. 2011 Apr;38(4):253-9. doi: 10.1097/OLQ.0b013e3181f70253. PMID 20966828
- [Background] Steinau M, Swan DC, Onyekwuluje JM, Brooks JT, Vellozzi C, Unger ER, The Sun Study Investigators. Differences and changes in human papillomavirus type 16 variant status in human immunodeficiency virus-positive adults are not uncommon. J Gen Virol. 2010 Aug;91(Pt 8):2068-2072. doi: 10.1099/vir.0.018663-0. Epub 2010 Apr 14. PMID 20392894
- [Background] Mondy KE, Gottdiener J, Overton ET, Henry K, Bush T, Conley L, Hammer J, Carpenter CC, Kojic E, Patel P, Brooks JT; SUN Study Investigators. High Prevalence of Echocardiographic Abnormalities among HIV-infected Persons in the Era of Highly Active Antiretroviral Therapy. Clin Infect Dis. 2011 Feb 1;52(3):378-86. doi: 10.1093/cid/ciq066. Epub 2010 Dec 9. PMID 21217185
- [Background] Dao CN, Patel P, Overton ET, Rhame F, Pals SL, Johnson C, Bush T, Brooks JT; Study to Understand the Natural History of HIV and AIDS in the Era of Effective Therapy (SUN) Investigators. Low vitamin D among HIV-infected adults: prevalence of and risk factors for low vitamin D Levels in a cohort of HIV-infected adults and comparison to prevalence among adults in the US general population. Clin Infect Dis. 2011 Feb 1;52(3):396-405. doi: 10.1093/cid/ciq158. PMID 21217186
- [Background] Kyser M, Buchacz K, Bush TJ, Conley LJ, Hammer J, Henry K, Kojic EM, Milam J, Overton ET, Wood KC, Brooks JT. Factors associated with non-adherence to antiretroviral therapy in the SUN study. AIDS Care. 2011 May;23(5):601-11. doi: 10.1080/09540121.2010.525603. PMID 21293992
- [Background] Overton ET, Patel P, Mondy K, Bush T, Conley L, Rhame F, Kojic EM, Hammer J, Henry K, Brooks JT; Sun Study Investigators. Cystatin C and baseline renal function among HIV-infected persons in the SUN Study. AIDS Res Hum Retroviruses. 2012 Feb;28(2):148-55. doi: 10.1089/AID.2011.0018. Epub 2011 May 25. PMID 21480819
- [Background] Mayer KH, Bush T, Henry K, Overton ET, Hammer J, Richardson J, Wood K, Conley L, Papp J, Caliendo AM, Patel P, Brooks JT; SUN Investigators. Ongoing sexually transmitted disease acquisition and risk-taking behavior among US HIV-infected patients in primary care: implications for prevention interventions. Sex Transm Dis. 2012 Jan;39(1):1-7. doi: 10.1097/OLQ.0b013e31823b1922. PMID 22183836
- [Background] Patel P, Bush T, Mayer KH, Desai S, Henry K, Overton ET, Conley L, Hammer J, Brooks JT; SUN Study Investigators. Prevalence and risk factors associated with herpes simplex virus-2 infection in a contemporary cohort of HIV-infected persons in the United States. Sex Transm Dis. 2012 Feb;39(2):154-60. doi: 10.1097/OLQ.0b013e318239d7fd. PMID 22249305
- [Background] Patel P, Bush T, Overton T, Baker J, Hammer J, Kojic E, Conley L, Henry K, Brooks JT; SUN Study Investigators. Effect of abacavir on acute changes in biomarkers associated with cardiovascular dysfunction. Antivir Ther. 2012;17(4):755-61. doi: 10.3851/IMP2020. Epub 2011 Dec 16. PMID 22301072
- [Background] Patel P, Bush T, Mayer K, Milam J, Richardson J, Hammer J, Henry K, Overton T, Conley L, Marks G, Brooks JT; SUN Study Investigators. Routine brief risk-reduction counseling with biannual STD testing reduces STD incidence among HIV-infected men who have sex with men in care. Sex Transm Dis. 2012 Jun;39(6):470-4. doi: 10.1097/OLQ.0b013e31824b3110. PMID 22592834
- [Background] Tedaldi EM, van den Berg-Wolf M, Richardson J, Patel P, Durham M, Hammer J, Henry K, Metzler S, Onen N, Conley L, Wood K, Brooks JT, Buchacz K; SUN Study Investigators. Sadness in the SUN: using computerized screening to analyze correlates of depression and adherence in HIV-infected adults in the United States. AIDS Patient Care STDS. 2012 Dec;26(12):718-29. doi: 10.1089/apc.2012.0132. PMID 23199190
- [Background] Baker JV, Hullsiek KH, Singh A, Wilson E, Henry K, Lichtenstein K, Onen N, Kojic E, Patel P, Brooks JT, Hodis HN, Budoff M, Sereti I; CDC SUN Study Investigators. Immunologic predictors of coronary artery calcium progression in a contemporary HIV cohort. AIDS. 2014 Mar 27;28(6):831-40. doi: 10.1097/QAD.0000000000000145. PMID 24370480
- [Background] Wilson EM, Singh A, Hullsiek KH, Gibson D, Henry WK, Lichtenstein K, Onen NF, Kojic E, Patel P, Brooks JT, Sereti I, Baker JV; Study to Understand the Natural History of HIV/AIDS in the Era of Effective Therapy (SUN Study) Investigators. Monocyte-activation phenotypes are associated with biomarkers of inflammation and coagulation in chronic HIV infection. J Infect Dis. 2014 Nov 1;210(9):1396-406. doi: 10.1093/infdis/jiu275. Epub 2014 May 9. PMID 24813472
- [Background] Escota GV, Patel P, Brooks JT, Bush T, Conley L, Baker J, Kojic EM, Hammer J, Onen NF; SUN Study Investigators. Short communication: The Veterans Aging Cohort Study Index is an effective tool to assess baseline frailty status in a contemporary cohort of HIV-infected persons. AIDS Res Hum Retroviruses. 2015 Mar;31(3):313-7. doi: 10.1089/AID.2014.0225. Epub 2015 Jan 20. PMID 25495766
- [Background] Battalora L, Buchacz K, Armon C, Overton ET, Hammer J, Patel P, Chmiel JS, Wood K, Bush TJ, Spear JR, Brooks JT, Young B; HIV Outpatient Study (HOPS) and SUN Study Investigators. Low bone mineral density and risk of incident fracture in HIV-infected adults. Antivir Ther. 2016;21(1):45-54. doi: 10.3851/IMP2979. Epub 2015 Jul 21. PMID 26194468